CLINICAL TRIAL: NCT02614326
Title: A Randomised Controlled Trial of the Efficacy of Autobiographical Memory Flexibility (MemFlex) Training in Preventing Relapse of Recurrent Depression
Brief Title: MemFlex to Prevent Depressive Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical Research Council Cognition and Brain Sciences Unit (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MemFlex to prevent relapse
Record Dates: First submitted 2015-11-19; First posted 2015-11-25 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Cognitive risk factors; Autobiographical memory; Cognitive bias; Relapse prevention
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memory Flexibility (MemFlex) Training (Experimental): MemFlex training draws on cognitive bias modification and memory specificity training techniques (Raes et al., 2009; Dalgleish et al., 2014). MemFlex is primarily self-guided and aims to reduce autobiographical memory biases associated with depression. The training is presented over one face-to-face session and eight self-guided sessions. In the initial session, the researcher introduces cued-recall tasks used throughout the workbook, and guides the participant in completion of the tasks. When understanding of the basic principles is satisfactory, the researcher assists the participant to set a schedule for completion of the workbook over the following four weeks. The participant will receive a phone call at the beginning of week three to check progress, and clarify any difficulties.
  Interventions: Behavioral: Autobiographical Memory Flexibility (MemFlex) training
- Psychoeducation (Placebo Comparator): The psychoeducation condition will also complete an initial face-to-face session. This session will cover the symptoms and causes of depression, and the workbook will be introduced. The workbook will consist of eight self-guided sessions that the individual will be required to complete over four weeks. The workbook content will cover the presentation of depression and basic information on factors associated with depression, such as worry, procrastination, and sleep difficulties. Each session consists of psychological theories of the topic, followed by a series of questions about the material to ensure participant engagement. The participant will receive a phone call from a team member at the beginning of week three to check progress, and clarify any difficulties.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Autobiographical Memory Flexibility (MemFlex) training — As in experimental arm description
  Other Names: MemFlex
  Arms: Memory Flexibility (MemFlex) Training
Behavioral: Psychoeducation — As in experimental arm description
  Arms: Psychoeducation

SUMMARY:
A wealth of research has demonstrated that they way in which the investigators recall our personal, autobiographical memories is influential in the course of depression. Biases in the recall of autobiographical memory occur in the midst of a depressive episode, and are shown to prolong symptoms, however these biases also remain when depression remits, and may predispose the individual towards relapse. A novel cognitive intervention, MemFlex, aims to train individuals to be flexible in their retrieval of autobiographical memories, and thereby reduce depressive relapse. Changes in memory bias may also have an effect on intermediate processes that increase risk of depression, such as rumination, impaired problem solving, and cognitive avoidance. This feasibility trial compares the effects of MemFlex and Psychoeducation in their ability to reduce memory bias and intermediate cognitive risk factors, and thereby depressive relapse, in individuals remitted from Major Depressive Disorder. Clinical outcome and process measures will be assessed immediately following completion of the intervention, at 6 months post-intervention, and at 12 months post-intervention. If encouraging, the results of this pilot trial may provide a foundation for a later phase trial.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for Major Depressive Disorder but is currently in remission, indexed on the Structured Clinical Interview for the DSM (SCID; First et al., 1996)
* 18 years of age or older

Exclusion Criteria:

* Meets criteria for a current Major Depressive Episode, indexed on the SCID
* Meets criteria for another mood disorder (e.g., Bipolar disorder), indexed on the SCID
* Current alcohol or substance dependence, or currently experiencing psychotic symptoms, indexed on the SCID
* Experience of intellectual disability, traumatic brain injury, or other neurological condition which may impact memory recall, assessed via self-report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-08 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Time to depressive relapse | 12 months post-intervention
  Length of time from post-intervention assessment to occurrence of any major depressive episode within the 12 month follow-up period
Number of depression free days at 12 month follow-up | 12 months post-intervention
  Number of depression free days as indexed by the Longitudinal Interval Follow-up Evaluation (Keller et al., 1987)

SECONDARY OUTCOMES:
Depressive status at 12 month follow-up | 12 months post-intervention
  Presence of a Major Depressive Episode as indexed by the Longitudinal Interval Follow-up Evaluation (Keller et al., 1987)
Depression symptoms at 12 month follow-up | 12 months post-intervention
  Score on the Beck Depression Inventory
Autobiographical memory retrieval | Measured within one week of completing the intervention
  Scores for specific and alternating blocks of the alternating instructions autobiographical memory task (Dritschel et al., 2013)

OTHER OUTCOMES:
Rumination | Measured within one week of completing the intervention, six months post-intervention and 12 months post-intervention
  Total and sub-scale scores on the Rumination Response Scale (Treynor, Gonzalez, Nolen-Hoeksema, 2003)
Problem solving | Measured within one week of completing the intervention, and six months post-intervention
  The total number of means and total effectiveness scores on the abbreviated version of the Means-Ends Problem Solving task (Marx, Williams, & Claridge, 1992)
Cognitive avoidance | Measured within one week of completing the intervention, six months post-intervention and 12 months post-intervention
  Total score on the Cognitive Avoidance Questionnaire (Sexton & Dugas, 2008)
Anxiety symptoms | Measured within one week of completing the intervention, six months post-intervention and 12 months post-intervention
  Total score on the Beck Anxiety Inventory (Beck & Steer, 1993)
Hopelessness | Measured within one week of completing the intervention, six months post-intervention and 12 months post-intervention
  Total score on the Beck Hopelessness Scale (Beck, Weissman, Lester, & Trexler, 1974)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Dalgleish, Principal Investigator — Medical Research Council Cognition and Brain Sciences Unit
Locations (2):
- United Kingdom (2):
  - MRC Cognition and Brain Sciences Unit, Cambridge
  - Cambridge and Peterborough NHS Foundation Trust, Cambridge

REFERENCES:
- [Background] Beck, A., Steer, R., & Brown, G. (1996). Manual for the Beck Depression Inventory II. San Antonio, TX: Psychological Corporation.
- [Background] Beck, A. T., & Steer, R. A. (1993). Beck Anxiety Inventory Manual. San Antonio, TX: Psychological Corporation.
- [Background] Dritschel B, Beltsos S, McClintock SM. An "alternating instructions" version of the Autobiographical Memory Test for assessing autobiographical memory specificity in non-clinical populations. Memory. 2014;22(8):881-9. doi: 10.1080/09658211.2013.839710. Epub 2013 Nov 12. PMID 24215524
- [Background] First, M. B., Spitzer, R. L., Gibbon, M., & Williams, J. B. (2002). Structured Clinical Interview for DSM-IV-TR Axis I Disorders, Research Version, Patient Edition. New York: Biometrics Research, New York State Psychiatric Institute.
- [Background] Treynor, W., Gonzalez, R., & Nolen-Hoeksema, S. (2003). Rumination reconsidered: A psychometric analysis. Cognitive Therapy and Research, 27, 247-259. doi: 10.1023/A:1023910315561
- [Background] Marx EM, Williams JM, Claridge GC. Depression and social problem solving. J Abnorm Psychol. 1992 Feb;101(1):78-86. doi: 10.1037//0021-843x.101.1.78. PMID 1537977
- [Background] Sexton KA, Dugas MJ. The Cognitive Avoidance Questionnaire: validation of the English translation. J Anxiety Disord. 2008;22(3):355-70. doi: 10.1016/j.janxdis.2007.04.005. Epub 2007 Apr 25. PMID 17544253
- [Background] Beck AT, Weissman A, Lester D, Trexler L. The measurement of pessimism: the hopelessness scale. J Consult Clin Psychol. 1974 Dec;42(6):861-5. doi: 10.1037/h0037562. No abstract available. PMID 4436473
- [Background] Keller MB, Lavori PW, Friedman B, Nielsen E, Endicott J, McDonald-Scott P, Andreasen NC. The Longitudinal Interval Follow-up Evaluation. A comprehensive method for assessing outcome in prospective longitudinal studies. Arch Gen Psychiatry. 1987 Jun;44(6):540-8. doi: 10.1001/archpsyc.1987.01800180050009. PMID 3579500
- [Derived] Hitchcock C, Gormley S, O'Leary C, Rodrigues E, Wright I, Griffiths K, Gillard J, Watson P, Hammond E, Werner-Seidler A, Dalgleish T. Study protocol for a randomised, controlled platform trial estimating the effect of autobiographical Memory Flexibility training (MemFlex) on relapse of recurrent major depressive disorder. BMJ Open. 2018 Jan 29;8(1):e018194. doi: 10.1136/bmjopen-2017-018194. PMID 29382674